CLINICAL TRIAL: NCT03750136
Title: HSS (Hypertonic Saline Solution) Plus High Dose Furosemide vs High Dose Furosemide in Nephrotic Syndrome - a Randomized Trial
Brief Title: Furosemide Alone or Unexpectedly With Solution of Hypertonic Saline in Nephrotic Syndrome
Acronym: FLUSH-NS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Principal Investigator, Alicja Rydzewska-Rosołowska, Principal Investigator, Medical University of Bialystok
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIKNT-001/2018
Record Dates: First submitted 2018-11-20; First posted 2018-11-21 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Nephrotic Syndrome
Keywords: diuretics
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Saline Solution, Hypertonic; Sodium Chloride; Furosemide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-dose furosemide & hypertonic saline (Experimental): furosemide i.v., 3% NaCl
  Interventions: Drug: Hypertonic saline; Drug: Furosemide Injection
- high-dose furosemide (Active Comparator): furosemide i.v.
  Interventions: Drug: Furosemide Injection

INTERVENTIONS:
Drug: Hypertonic saline — high dose furosemide with hypertonic saline 3x daily
  Other Names: 3% saline
  Arms: high-dose furosemide & hypertonic saline
Drug: Furosemide Injection — high dose furosemide

SUMMARY:
The trial will test the hypothesis that hypertonic saline on top of standard diuretic treatment will help achieve adequate diuresis in patients with nephrotic syndrome.

DETAILED DESCRIPTION:
Objectives:

Edema is one of the major clinical manifestations of nephrotic syndrome. All patients are initially treated with diuretics and sodium restriction but the results are sometimes not satisfactory. Hypertonic saline solutions have been studied in congestive heart failure and a meta-analysis confirmed it's role in achieving adequate diuresis and protecting patients against acute kidney injury although the proposed mechanism of action is not known (osmotic action?, inhibition of renin-angiotensin-aldostrerone system?, increase in renal perfusion?, myocardial contractility?). The investigators therefore hypothesized that it may exert beneficial effects also in nephrotic syndrome.

Treatment protocol:

A prospective placebo-controlled randomized trial. Subjects will be randomized to high-dose furosemide vs high-dose furosemide plus hypertonic intravenous saline in a 1:1 fashion. All subjects will receive furosemide tid (starting with 3x40 mg i.v.) with or without hypertonic saline solution (3x100 ml of 3% NaCl - in a combined infusion lasting 10 minutes). Subjects randomized to furosemide only will receive 3x100 ml of 5% glucose (in a combined infusion lasting 10 minutes). The dose of furosemide will be determined by the investigator based on patients weight, severity of edema, 24-h urine volume, kidney function. In case of poor clinical response (urine volume below 1000 ml) the investigator will be able to titrate the furosemide dose up to 3x180 mg i.v. All patients will be kept on low-salt diet and water restriction (500-1000 ml/day), their weight will assessed every morning before breakfast and measurement of 24-h urine volume will be performed every day. Additionally BNP levels will be measured at baseline and after 5 days of treatment. Treatment will be continued for 5 days. The primary measure of efficacy will be urine volume and the rate of acute kidney injury (AKI), secondary measure of efficacy will be the expected decrease in brain natriuretic peptides (BNP) levels and the length of hospitalization.

Hydrochlorothiazide, spironolactone and other diuretics use will be contraindicated during the study. Patients will be required to receive standard concurrent therapy as determined by their attending physician and according to current guidelines (including steroids and other immunosuppresives).

ELIGIBILITY:
Inclusion Criteria:

* 30 consecutive patients with nephrotic syndrome (proteinuria over 3.5 g/day, edema, hypoalbuminemia, dysproteinemia) admitted to II Nephrology Department from November 2018 onwards within 48h of admission,
* age above 18,
* informed consent.

Exclusion Criteria:

* AKI (acute kidney injury) - AKIN criteria level 3,
* CKD (chronic kidney disease) stage 4 and 5 according to KDIGO (Kidney Disease: Improving Global Outcomes),
* concomittant heart failure NYHA (New York Heart Association) class III or worse,
* active liver disease and liver failure,
* terminal neoplastic disease,
* serum sodium above 145 mmol/l,
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12-15 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Diuresis | 5 days
  ml of diuresis

SECONDARY OUTCOMES:
Length of hospitalisation | 14 days
  days
BNP levels | 5 days
  pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Alicja Rydzewska-Rosolowska, MD, Principal Investigator — Medical University of Białystok
Locations (1):
- II Department of Nephrology and Hypertension, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Licata G, Di Pasquale P, Parrinello G, Cardinale A, Scandurra A, Follone G, Argano C, Tuttolomondo A, Paterna S. Effects of high-dose furosemide and small-volume hypertonic saline solution infusion in comparison with a high dose of furosemide as bolus in refractory congestive heart failure: long-term effects. Am Heart J. 2003 Mar;145(3):459-66. doi: 10.1067/mhj.2003.166. PMID 12660669
- [Background] Paterna S, Parrinello G, Amato P, Dominguez L, Pinto A, Maniscalchi T, Cardinale A, Licata A, Amato V, Licata G, Di Pasquale P. Tolerability and efficacy of high-dose furosemide and small-volume hypertonic saline solution in refractory congestive heart failure. Adv Ther. 1999 Sep-Oct;16(5):219-28. PMID 10915397
- [Background] Paterna S, Di Pasquale P, Parrinello G, Amato P, Cardinale A, Follone G, Giubilato A, Licata G. Effects of high-dose furosemide and small-volume hypertonic saline solution infusion in comparison with a high dose of furosemide as a bolus, in refractory congestive heart failure. Eur J Heart Fail. 2000 Sep;2(3):305-13. doi: 10.1016/s1388-9842(00)00094-5. PMID 10938493